CLINICAL TRIAL: NCT04704258
Title: Clinical Study of a Novel Transcatheter Anti-embolic Filter (FLOWer) for Cerebral Protection During Aortic Valve Interventions
Brief Title: NAUTILUS CE-mark Trial of the FLOWer Cerebral Embolic Protection Device
Acronym: NAUTILUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AorticLab Srl (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #2020-01 (EU)
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Aortic Valve Stenosis; Intracranial Embolism and Thrombosis
Keywords: TAVI; Transcatheter Anti-embolic Filter; Cerebral Embolic Protection; Embolic Protection Device; Debris; Embolic material
MeSH Terms: conditions — Aortic Valve Stenosis; Intracranial Embolism and Thrombosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVI + Embolic protection (Experimental): Subjects with severe native aortic valve stenosis who meet the clinically approved indications for aortic valve interventions such as TAVI
  Interventions: Procedure: TAVI (Transcatheter Aortic Valve Implant); Device: FLOWer Embolic Protection System

INTERVENTIONS:
Procedure: TAVI (Transcatheter Aortic Valve Implant) — Placement of a filter to capture and remove emboli or debris detached during any transcatheter heart procedures
Device: FLOWer Embolic Protection System — FLOWer Embolic Protection System
  Other Names: transcatheter embolic protection for TAVI procedures

SUMMARY:
The purpose of this clinical study is to assess the safety, performance, and treatment effect of the use of the AorticLab FLOWer System, in preventing cerebral thromboembolic complications in patients with indication for a TAVI (Transcatheter Aortic Valve Implant).

DETAILED DESCRIPTION:
A single arm, prospective, multicenter non-randomized clinical study of the AorticLab FLOWer System to prevent embolic complications during transcatheter aortic valve procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age ≥ 18 years
2. Subject is scheduled to undergo transfemoral aortic valve implant (TAVI) procedure on a stenotic native aortic valve and is qualified based on pre-operative CT-scan examination (trans-thoracic echocardiogram (TTE) can be used as confirmatory assessment)
3. Subject anatomy with Ilio-femoral artery segment compatible with a 12 F device catheter size
4. The subject and the treating physician agree that the subject will undergo the scheduled pre-procedural testing and return for all required post-procedure follow-up visits
5. The subject, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (EC) or Institutional Review Board (IRB)

Exclusion Criteria:

Clinical exclusion criteria (preoperative screening)

1. Subjects with hypercoagulable state that cannot be corrected by additional periprocedural heparin
2. Subjects with contraindication to cerebral MRI
3. Subjects with a history of a stroke or transient ischemic attack within the prior 6 months
4. Subjects with known diagnosis of acute myocardial infarction (AMI) within 30 days preceding the index procedure
5. Renal insufficiency (creatinine > 3.0 mg/dL or Glomerular Filtration Rate GFR < 30) and/or renal replacement therapy at the time of screening
6. Subjects with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, patients who will refuse transfusion, or patients with an active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 3 months
7. Subjects with known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated
8. Subject is currently participating in another drug or device clinical study or has other medical illnesses that may cause the subject to be non-compliant with the protocol or confound the data interpretation
9. Subjects with a previously implanted prosthetic aortic valve (i.e., planned valve-in-valve with a TAVI)
10. Subject requires an emergent procedure
11. Subject has active major psychiatric disease
12. Subjects with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
13. Subject has an ejection fraction of 30% or less
14. Subjects with active endocarditis or other systemic infection
15. Subjects undergoing therapeutic thrombolysis
16. Subject is pregnant or lactating. Pregnancy confirmed by positive urine or serum test

Computerized Tomographic exclusion criteria (preoperative screening)

1. Subjects with documented friable or mobile atherosclerotic plaque in the aortic arch
2. Subjects with echocardiographic evidence of aortic mass, thrombus or vegetation
3. Subjects with a diameter of the ascending aorta < 25 and > 39 mm at baseline CT (measured 10 mm upstream of the first vessel of the brachiocephalic trunk)
4. Subjects undergoing transcatheter aortic valve implantation (TAVI) via the trans-axillary, trans-subclavian, or trans-aortic route
5. Subjects with severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery of sheath vascular access
6. Subjects in whom the aortic arch is heavily calcified, severely atheromatous, or severely tortuous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
FLOWer Device Safety: Rate of Major Adverse Cardiac and Cerebrovascular Events | 30 days
  Primary Safety Endpoint: FLOWer device Safety, rate of Major Adverse Cardiac and Cerebrovascular Events (MACCEs) related to FLOWer device and procedure as adjudicated by a Clinical Event Committee. MACCEs are based on the Valve Academic Research Consortium (VARC- 3) criteria:
  * all death;
  * all stroke (disabling and non-disabling);
  * acute kidney injury (stage 3 at discharge or 72 hours post index procedure, whichever occurs first)
Reduction in total volume of new cerebral lesions in all territories at serial DWMRI | Within 2-5 days after procedure vs. baseline
  Primary Clinical Benefit Endpoint: Reduction in total volume of new cerebral lesions in all territories at serial DWMRI, compared to historical data in control arm (unprotected) data from previous randomized studies

SECONDARY OUTCOMES:
Cumulative occurrence of Serious Clinical Events related to FLOWer device and procedure as adjudicated by a Clinical Event Committee. | 7 and 30 days
  Secondary Safety Endpoint: Cumulative occurrence of Serious Clinical Events related to FLOWer device and procedure as adjudicated by a Clinical Event Committee. all-cause mortality including cardiovascular mortality;
  * all stroke (disabling and non-disabling);
  * bleeding (life-threatening or disabling);
  * acute kidney injury (stage 3 at discharge or 72 hours post index procedure, whichever occurs first);
  * major device access related vascular complications;
  * coronary artery obstruction requiring intervention;
  * valve-related dysfunction requiring repeat procedure (balloon aortic valvuloplasty, repeat TAVI, or surgical aortic valve replacement).
Brain imaging (DW-MRI) | Within 2-5 days after procedure vs. baseline
  Secondary Clinical Benefit Endpoints: Acute cerebral embolic burden reduction after TAVI, defined as number and volume of new cerebral lesions in all cerebral territories assessed by DW-MRI
Neurocognitive | 2-7 days and 30-days vs. baseline
  Secondary Clinical Benefit Endpoints: Neurocognitive protection assessed by NIHSS, Montreal Cognitive Assessment, and mRS
Technical Success | Immediately after procedure
  Secondary Performance Endpoints: Technical Success defined as successful placement, insertion and removal of the FLOWer System
Debris capture | Immediately after procedure
  Secondary Performance Endpoints: Debris captured by the FLOWer System with gross and histopathological evaluation including particle size and composition
FLOWer System Usability | Immediately after procedure
  Secondary Performance Endpoints: FLOWer System Usability graded by the Investigator with a 5-point Likert scale
  The minimum and the maximum values of the scale are defined as follows:
  (1) Unacceptable; (2) Poor; (3) Acceptable; (4) Good; (5) Excellent

CONTACTS AND LOCATIONS:
Overall Officials: Franco Osta, Study Chair — AorticLab Srl
Locations (8):
- Belgium (2):
  - HartCentrum, Ziekenhuis Netwerk Antwerpen (ZNA) Middelheim, Antwerp
  - CUB Hôpital Erasme (ULB), Brussels
- Italy (6):
  - Casa di Cura Policlinico di Monza, Monza, MB
  - IRCCS Ospedale San Raffaele, Milan, MI
  - IRCCS Policlinico San Donato, San Donato Milanese, MI
  - San Carlo Azienda Ospedaliera Regionale, Potenza, PZ
  - Centro Cardiologico Monzino IRCCS, Milan
  - Clinica San Gaudenzio, Novara

REFERENCES:
- See also: Aorticlab Sponsor website — http://www.aorticlab.ch
- See also: Meditrial Clinical Research Organization — http://www.meditrial.net